CLINICAL TRIAL: NCT04026503
Title: The Live Long Walk Strong Rehabilitation Program: What Features Improve Mobility Skills?
Brief Title: Live Long Walk Strong (LLWS) Rehabilitation Program: What Features Improve Mobility Skills
Acronym: LLWS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E3095-R
Record Dates: First submitted 2019-07-18; First posted 2019-07-19 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Mobility Limitation
Keywords: Rehabilitation; Aging; Mobility Skills
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Intervention Model Description: Participants are assigned to 8 week Live Long Walk Strong rehabilitation or 8 week wait list control then the LLWS rehabilitation program.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants are randomized through block permuted generated lists performed by the study biostatistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Live Long Walk Strong (Experimental): 8 week rehabilitation program
  Interventions: Other: Live Long Walk Strong rehabilitation program
- 8 week wait list control (Active Comparator): 8 week wait list then followed by 8 weeks of the Live Long Walk Strong rehabilitation program
  Interventions: Other: Live Long Walk Strong rehabilitation program

INTERVENTIONS:
Other: Live Long Walk Strong rehabilitation program — Live Long Walk Strong is a rehabilitation program that focuses on impairments known to contribute to mobility decline that are not considered standard of care in rehab and addresses behavioral change within the context of rehabilitation.

SUMMARY:
This study is being performed to evaluate the efficacy of the Live Long Walk Strong rehabilitation program in Veterans 50 years and older. This study will also examine the features of the program that contribute to improved gait speed.

DETAILED DESCRIPTION:
Due to COVID-19, currently completed a virtual version of the LLWS intervention study.

The investigators are currently recruiting for the original study design in-person.

This study is a 4 year phase II randomized clinical trial study design. This study will provide important information about the mechanisms that contribute to meaningful improvement in mobility, the benefits of a novel mode of physical therapy care, and the duration of treatment effect.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Aged 50 and older
* Community dwelling
* Ability to speak and understand English
* Usual gait speed 0.5 m/s- 1.0 m/s Activity modifications and access to telehealth rehabilitation

Exclusion Criteria:

* Presence of a terminal disease
* A major medical problem, unstable chronic condition, or psychiatric disorder that interferes with safe and successful testing and training
* Myocardial infarction or major surgery in previous 3 months
* Planned major surgery
* Baseline short physical performance battery score less than 4
* Use of a walker
* Modified mini mental status examination score less than or equal to 77
* Presence of a significant disease specific impairment such as:

  * peripheral neurologic impairment
  * orthopedic impairment
  * visual impairment

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-11-07 (Actual)

PRIMARY OUTCOMES:
Gait Speed | within 2 weeks, 8 weeks, 16 weeks follow up
  Gait speed change will be assessed within 2 weeks post intervention and then in 8 and 16 weeks of subsequent follow-up.
  Virtual only pilot assessing the feasibility of the LLWS program in a virtual format.

SECONDARY OUTCOMES:
Lower Extremity Power | within 2 weeks, 8 weeks, 16 weeks follow up
  Lower extremity power measure will be assessed at 3 time points post intervention. Power will be assessed via a keiser machine (force) and stair climb test (seconds).
Trunk Muscle Endurance | within 2 weeks, 8 weeks, 16 weeks follow up
  Trunk muscle endurance will be measured at 3 time points post intervention. Trunk endurance will be assessed via saunders table through time (seconds) held in a fixed position.
Gait Variability | within 2 weeks, 8 weeks, 16 weeks follow up
  Gait variability will be measured at 3 time points post intervention. Gait variability will be assessed via zeno gait mat measurement of step length, step width and other measures of gait quality captured via the pkmas software within the zeno gait mat.

OTHER OUTCOMES:
Cognition | Within 2 weeks of intervention end
  A cognitive battery, including the DKEFS verbal fluency and DKEFS trail making tests will be assessed pre and post intervention (within 2 weeks). For all tests both scaled scores (1-19) will be reported. For DKEFS trail making tests raw scores will also be reported.
Adherence | Within 2 weeks of intervention end
  Adherence will be assessed by drop out status from the study between enrollment and the first follow up visit (2 weeks post intervention), defined as a yes or no status.
Compliance | 16 weeks follow up
  Compliance with be assessed separately by the number of intervention sessions attended (out of 10) and the number of reported exercise days during follow up period (over 16-week time period).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan F. Bean, MD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wingood M, Linsky AM, Harris R, Bamonti P, Moye J, Bean JF. Research Protocol Adaptations During the COVID-19 Pandemic: A Process Evaluation. J Aging Phys Act. 2023 Sep 12;32(1):62-68. doi: 10.1123/japa.2023-0052. Print 2024 Feb 1. PMID 37699586
- [Background] Harris R, Brach JS, Moye J, Ogawa E, Ward R, Halasz I, Bean J. The Live Long Walk Strong Rehabilitation Program Study: Design and Methods. Arch Rehabil Res Clin Transl. 2022 May 29;4(3):100205. doi: 10.1016/j.arrct.2022.100205. eCollection 2022 Sep. PMID 36123980
- [Background] Bamonti PM, Moye J, Harris R, Kallmi S, Kelly CA, Middleton A, Bean JF. Development of a Coaching Protocol to Enhance Self-efficacy Within Outpatient Physical Therapy. Arch Rehabil Res Clin Transl. 2022 Apr 21;4(2):100198. doi: 10.1016/j.arrct.2022.100198. eCollection 2022 Jun. PMID 35756988
- [Result] Harris R, Ogawa EF, Ward RE, Fitzelle-Jones E, Travison T, Brach JS, Bean JF. Feasibility and Preliminary Efficacy of Virtual Rehabilitation for Middle and Older Aged Veterans With Mobility Limitations: A Pilot Study. Arch Rehabil Res Clin Transl. 2024 Feb 12;6(2):100325. doi: 10.1016/j.arrct.2024.100325. eCollection 2024 Jun. PMID 39006121
- [Result] Ganguly A, Hampton T. Calcium-dependence of serotonin-mediated aldosterone secretion and differential effects of calcium antagonists. Life Sci. 1985 Apr 15;36(15):1459-64. doi: 10.1016/0024-3205(85)90053-0. PMID 3982220
- [Result] Ogawa EF, Harris R, Moye J, Bean JF, Kim B. Veterans' Motivation, Preference, and Feedback After Completing a Novel Physical Therapy Treatment. J Aging Phys Act. 2025 Jan 17;33(4):379-386. doi: 10.1123/japa.2023-0446. Print 2025 Aug 1. PMID 39826533

DOCUMENTS (1):
  • Informed Consent Form (2021-01-04): https://cdn.clinicaltrials.gov/large-docs/03/NCT04026503/ICF_000.pdf